CLINICAL TRIAL: NCT02333435
Title: Étude randomisée, contrôlée, de Phase II, Effets d'un Supplement d'oméga-3 (EPA) Sur l'Inflammation, la prolifération Cellulaire et la qualité de Vie Chez Des Patients Avec Cancer de la Prostate traités Par Prostatectomie Radicale
Brief Title: Effects of EPA on Prostate Cancer Cells Proliferation and Quality of Life
Acronym: RCT-EPA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-1012
Record Dates: First submitted 2014-12-17; First posted 2015-01-07 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Omega-3 fatty acids; Quality of life; inflammation; cellular proliferation
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation; Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Purified EPA group (Experimental): 3g per day of purified EPA, capsules, to be taken once a day, for 14 months.
  Interventions: Dietary Supplement: EPA
- Placebo group (Experimental): 3 g per day of high-oleic sunflower oil capsules, to be taken once a day, for 14 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: EPA — 3g/day of purified EPA , capsules, taken once daily, for 14 months
  Arms: Purified EPA group
Dietary Supplement: Placebo — 3g/day of placebo (high oleic sunflower oil) , capsules, taken once daily, for 14 months
  Other Names: High oleic sunflower oil
  Arms: Placebo group

SUMMARY:
Prostate cancer, the most frequently diagnosed cancer among occidental men, is associated with a major individual and societal burden. Although still controversial, the literature suggests that a high consumption of omega-3 fatty acids (ω3) has protective effects against prostate cancer. One of the proposed mechanisms of action of ω3 lies in their anti-inflammatory properties. In addition, there are some observational evidences suggesting an association of ω3 intake with a lower rate of depression in cancer patients. However, no clinical study has tested the efficacy of ω3 supplementation on psychological and quality of life outcomes in that population. Several evidences point to a possible involvement of inflammation in psychological issues. Reducing the systemic inflammatory state may have beneficial impact on the quality of life of these patients. Preliminary work from this team of investigators, in a cohort of patients managed with active surveillance for their low-grade prostate cancer, show a strong inverse association between the risk of prostate cancer progression (to high-grade) and the level of prostatic eicosapentanoic acid (EPA- a type of ω3).

HYPOTHESIS: EPA-rich monoglycerides fish oil (MAG-EPA) has global positive effects on prostate cancer cell proliferation, inflammation and on the patient's psychosocial functioning and quality of life.

The investigators propose a double blind, randomized controlled clinical trial. 130 consecutive patients suffering from high-risk prostate cancer who choose to be treated by radical prostatectomy will be eligible to this study. The presence of high-grade cancer will be mandatory.

The intervention, a daily supplementation with 3g supplement of fish oil monoglycerides rich in EPA, vs. placebo capsules containing high oleic sunflower oil, will start six weeks before the prostatectomy and will continue for one year after surgery. The potential confounding variables will be measured before the start of the intervention: age, anthropometric parameters, stage and clinical and pathological tumor grade (Gleason score), pre-operative level of prostate specific antigen and diet.

This project proposes a simple intervention by dietary supplementation that could eventually help to reduce the incidence and/or progression of prostate cancer, and the consequences of its treatment, and thus could contribute to diminish the heavy individual and societal burden of prostate cancer. The clinical data generated by this trial will serve as solid basis for a large-scale phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer (Gleason score >= 7)
* Patient has chosen to undergo radical prostatectomy
* Patient agrees to stop taking any omega-3 supplements at least 3 months before the start of the study
* Patient has provided informed consent

Exclusion Criteria:

* Allergy to fish and sunflower
* Suffering from a bipolar disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Prostate Cancer Proliferative Index | 6 weeks
  At 6 weeks post study entry, the prostate of the patient will be removed by prostatectomy. The tissue will be preserved in paraffin blocks. The tumour will be identified and the level of Ki-67 in the tumour will be quantified.

SECONDARY OUTCOMES:
Change in Inflammatory mediators levels- Systemic | 6 weeks, 1 year
  The changes in levels of systemic inflammatory mediators, relative to their baseline levels, at the time of radical prostatectomy and at one year post-radical prostatectomy, will be measured. The levels of mediators will be expressed in pg/mL and quantified using validated techniques.
Modulation of Inflammatory mediators levels - Prostatic | 6 weeks, 1 year
  The differences in the levels of expression of inflammatory mediators between both treatment groups will be measured in the peripheral zone of the prostate before surgical prostate dissection/ischemia. The levels of mediators will be expressed in pg/mL and quantified using validated techniques. Further validation could be performed using immunohistochemistry techniques.
Modulation of the Quality of life of patients | 6 weeks, 3, 6, 9 and 12 months post radical prostatectomy
  Validated questionnaires will be used to measure the modulation of the treatment on Quality of Life of the patients, which will include questions on mood, anxiety levels, sleep and cognition.
Modulation of the psychosocial functioning of patients | 6 weeks, 3, 6, 9 and 12 months post radical prostatectomy
  Validated questionnaires will be used to measure the modulation of the treatment on psychosocial functioning of the patients, which will include questions on mood, anxiety levels, sleep and cognition.
Impact of inflammation on Quality of life | 6 weeks, 3, 6, 9 and 12 months post radical prostatectomy
  The impact of changes in inflammatory mediators levels induced by EPA supplementation on quality of life scores will be measured. To do so, we will use appropriate and powerful statistical tests.
Impact of inflammation on psychosocial functioning | 6 weeks, 3, 6, 9 and 12 months post radical prostatectomy
  The impact of changes in inflammatory mediators levels induced by EPA supplementation and changes in psychosocial functioning scores will be measured. To do so, we will use appropriate and powerful statistical tests.

OTHER OUTCOMES:
Fatty acid profiles in red blood cell membranes, change relative to baseline | 6 weeks, 3, 6, 9, 12 months post radical prostatectomy
  The difference of fatty acid levels between both groups, relative to baseline, will be quantified using gas chromatography coupled with mass spectrometry and expressed as relative percentages of total fatty acids.
Fatty acid profiles in prostate tissue | 6 weeks
  The difference of fatty acid levels between both groups at prostatectomy will be quantified using gas chromatography coupled with mass spectrometry and expressed as relative percentages of total fatty acids, and in absolute level (mg per gram of tissue).
Impact of EPA supplementation on radical prostatectomy complications | 6 weeks
  The difference in perioperative bleeding, laboratory tests (hemoglobin, hematocrit and platelets) and surgical complications between both group will be examined at surgery.
Impact of EPA supplementation on cancer aggressiveness | 6 weeks
  Pathological reclassification of cancer grade (ISUP grading system) and stage between the prostate diagnostic biopsy and the prostatectomy specimen will be compared between both groups.
Change on PSA level (ng/mL), relative to baseline | 6 weeks, 3, 6, 9 and 12 months post radical prostatectomy
  PSA change relative to baseline will be measured for both groups.
Impact of EPA supplementation on biochemical recurrence | 5 years post radical prostatectomy
  The biochemical recurrence, defined as a PSA level ≥ 0.2 ng/mL after reaching a non-detectable level at three months post-surgery, will be evaluated for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fradet, MD, PhD, Principal Investigator — Laval University and Hotel Dieu-de-Quebec
Locations (1):
- Centre de Recherche Clinique et Evaluative en Oncologie - Hotel Dieu de Quebec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Robitaille K, Guertin MH, Jamshidi A, Xu HW, Hovington H, Pelletier JF, Beaudoin L, Gevariya N, Lacombe L, Tiguert R, Caumartin Y, Dujardin T, Toren P, Lodde M, Racine E, Trudel D, Perigny M, Duchesne T, Savard J, Julien P, Fradet Y, Fradet V. A phase IIb randomized placebo-controlled trial testing the effect of MAG-EPA long-chain omega-3 fatty acid dietary supplement on prostate cancer proliferation. Commun Med (Lond). 2024 Mar 22;4(1):56. doi: 10.1038/s43856-024-00456-4. PMID 38519581
- [Derived] Savard J, Moussa H, Pelletier JF, Julien P, Lacombe L, Tiguert R, Caumartin Y, Dujardin T, Toren P, Pouliot F, Lodde M, Fradet Y, Robitaille K, Fradet V. Effects of omega-3 supplementation on psychological symptoms in men with prostate cancer: Secondary analysis of a double-blind placebo-controlled randomized trial. Cancer Med. 2023 Oct;12(19):20163-20176. doi: 10.1002/cam4.6598. Epub 2023 Oct 3. PMID 37787025
- [Derived] Guertin MH, Robitaille K, Pelletier JF, Duchesne T, Julien P, Savard J, Bairati I, Fradet V. Effects of concentrated long-chain omega-3 polyunsaturated fatty acid supplementation before radical prostatectomy on prostate cancer proliferation, inflammation, and quality of life: study protocol for a phase IIb, randomized, double-blind, placebo-controlled trial. BMC Cancer. 2018 Jan 10;18(1):64. doi: 10.1186/s12885-017-3979-9. PMID 29321047